CLINICAL TRIAL: NCT01838681
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Flexible-dose Long-term Study to Evaluate the Maintenance of Efficacy and Safety of 1 to 3 mg/Day of Brexpiprazole as Adjunctive Treatment in Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Brief Title: Brexpiprazole as Adjunctive Treatment in Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14570A; 2012-001380-76 (EudraCT Number)
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Interventions: Drug: Placebo; Drug: ADT
- Brexpiprazole (Experimental): Brexpiprazole adjunct to open-label treatment with a commercially available ADT
  Interventions: Drug: Brexpiprazole; Drug: ADT

INTERVENTIONS:
Drug: Placebo — Once daily, tablets, orally
  Arms: Placebo
Drug: Brexpiprazole — 1, 2, or 3 mg/day, once daily dose, tablets, orally. Uptitration in weekly steps from 1 mg/day
  Arms: Brexpiprazole
Drug: ADT — Duloxetine, escitalopram, fluoxetine, paroxetine IR, sertraline, venlafaxine XR; dosing according to label

SUMMARY:
To evaluate the long-term efficacy and safety of brexpiprazole as an adjunctive treatment to an antidepressant treatment (ADT) for adult patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
The total duration of the study was 32 weeks and the study consisted of Periods A, B, and A+. Patients entered the study in Period A and were treated open-label with one of six commercially available antidepressant treatments (ADTs) for 8 weeks. Patients who met the blinded response criteria at the Week 6 Visit, were deemed early responders and were withdrawn from the study. At Week 8, patients with inadequate response to placebo + ADT, as per the randomisation criteria, entered Period B and were randomised to received double-blind brexpiprazole + ADT or placebo + ADT for 24 weeks. Non-randomised patients continued in Period A+ and received placebo + ADT until the end of the study. The primary objective was to compare the efficacy and safety of brexpiprazole with placebo. This comparison occurred Period B; therefore, the focus is Period B.

ELIGIBILITY:
Inclusion Criteria:

* The patient is an outpatient consulting a psychiatrist.
* The patient has an MDD diagnosed according to DSM-IV-TR™. The current Major Depressive Episode (MDE) should be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has a moderate to severe depression and an insufficient response to at least one and no more than three adequate antidepressant treatments.
* The patient agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

* The patient has any current psychiatric disorder or Axis I disorder (DSM-IV-TR™ criteria), established as the primary diagnosis, other than MDD.
* The patient has a current Axis II (DSM-IV-TR™) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypical or histrionic personality disorder.
* The patient has experienced/experiences hallucinations, delusions or any psychotic symptomatology in the current MDE.
* The patient suffers from mental retardation, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient, in the opinion of the investigator or according to Columbia-Suicide Severity Rating Scale (C-SSRS), is at significant risk of suicide.
* The patient has had neuroleptic malignant syndrome.
* The patient has any relevant medical history or current presence of systemic disease.
* The patient has, at the Screening Visit an abnormal ECG that is, in the investigator's opinion, clinically significant.
* The patient has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, that has not been in remission for >5 years prior to the first dose of IMP.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1986 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (107):
- United States (8):
  - US041, Little Rock, Arkansas
  - US043, Cerritos, California
  - US042, Temecula, California
  - US053, Flowood, Mississippi
  - US040, Brooklyn, New York
  - US046, Houston, Texas
  - US052, Houston, Texas
  - US047, Milwaukee, Wisconsin
- Bulgaria (7):
  - BG007, Kardzhali
  - BG002, Pazardzhik
  - BG003, Rousse
  - BG001, Sofia
  - BG004, Sofia
  - BG005, Varna
  - BG006, Varna
- Canada (5):
  - CA003, Burlington
  - CA004, Edmonton, Alberta
  - CA001, Kingston
  - CA002, Montral
  - CA005, Montreal
- Estonia (6):
  - EE002, Tallinn
  - EE003, Tallinn
  - EE006, Tallinn
  - EE001, Tartu
  - EE005, Tartu
  - EE004, Võru
- Finland (6):
  - FI002, Helsinki
  - FI003, Helsinki
  - FI006, Helsinki
  - FI001, Kuopio
  - FI007, Pori
  - FI009, Tampere
- Germany (14):
  - DE007, Berlin
  - DE014, Berlin
  - DE015, Berlin
  - DE006, Bielefeld
  - DE010, Bochum
  - DE012, Gelsenkirchen
  - DE009, Hanover
  - DE022, Hattingen
  - DE008, Heidelberg
  - DE017, Leipzig
  - DE001, Nuremberg
  - DE004, Nuremberg
  - DE002, Schwerin
  - DE016, Wiesbaden
- Latvia (5):
  - LV004, Daugavpils
  - LV005, Jelgava
  - LV002, Liepāja
  - LV003, Riga
  - LV001, Strenči
- Lithuania (6):
  - LT003, Kaunas
  - LT006, Kaunas Region
  - LT001, Palanga
  - LT005, Šilutė
  - LT002, Vilnius
  - LT004, Vilnius
- Mexico (4):
  - MX009, Guadalajara
  - MX008, León
  - MX002, Monterrey
  - MX003, Monterrey, Nuevo Len
- Poland (13):
  - PL010, Bialystok
  - PL016, Bialystok
  - PL017, Bydgoszcz
  - PL007, Chełmno
  - PL002, Gdansk
  - PL011, Gorlice
  - PL018, Kielce
  - PL013, Leszno
  - PL001, Lublin
  - PL006, Lublin
  - PL014, Szczecin
  - PL012, Torun
  - PL019, Torun
- Romania (4):
  - RO003, Bucharest
  - RO006, Bucharest
  - RO001, Iași
  - RO004, Timișoara
- Russia (9):
  - RU002, Moscow
  - RU004, Moscow
  - RU003, Saint Petersburg
  - RU006, Saint Petersburg
  - RU007, Saint Petersburg
  - RU010, Saint Petersburg
  - RU014, Saint Petersburg
  - RU012, Saratov
  - RU005, Stavropol
- South Korea (2):
  - KR001, Seoul
  - KR004, Seoul
- Sweden (4):
  - SE008, Halmstad
  - SE006, Malmo
  - SE009, Skövde
  - SE001, Stockholm
- Ukraine (8):
  - UA006, Kharkiv
  - UA007, Kherson,Vil. Stepanivka
  - UA003, Kiev
  - UA014, Kiev
  - UA002, Kyiv
  - UA005, Lviv
  - UA012, Ternopil
  - UA009, Vinnytsia
- United Kingdom (6):
  - GB003, Blackpool
  - GB005, Bognor Regis
  - GB002, Bradford
  - GB004, Cannock
  - GB001, Leeds
  - GB006, Winwick

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1986 patients were enrolled; 1982 received open-label ADT plus double-blind placebo in the 8-week Period A. In the 24-week Period B, 886 patients were randomised and 885 were treated with open-label ADT plus double-blind brexpiprazole or placebo. Non-randomised patients continued in Period A+ and received open-label ADT plus double-blind placebo.
Groups:
- Period A Placebo and ADT (8 Weeks): Placebo adjunct to open-label treatment with ADT
  Placebo: Once daily, tablets, orally
- Period B Placebo and ADT (24 Weeks Randomised Treatment); Period A+ Placebo and ADT (Non-randomised Patients): Placebo adjunct to open-label treatment with ADT (same ADT as in Period A)
  Placebo: Once daily, tablets, orally
- Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment): Brexpiprazole adjunct to open-label treatment with ADT (same ADT as in Period A)
  Brexpiprazole: flexible dose; 1, 2, or 3 mg/day, once daily, tablets, orally
Period: Period A
Arm/Group | Period A Placebo and ADT (8 Weeks) | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment) | Period A+ Placebo and ADT (Non-randomised Patients)
Started | 1986 | 0 | 0 | 0
Completed | 1661 | 0 | 0 | 0
Not Completed | 325 | 0 | 0 | 0
Not completed — Adverse Event | 39 | 0 | 0 | 0
Not completed — Lack of Efficacy | 21 | 0 | 0 | 0
Not completed — Early response | 148 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 70 | 0 | 0 | 0
Not completed — Protocol Violation | 16 | 0 | 0 | 0
Not completed — Non-compliance with IMP | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0
Not completed — Withdrawal before treatment | 4 | 0 | 0 | 0
Not completed — Administrative or other reasons | 17 | 0 | 0 | 0
Period: Period B/A+
Arm/Group | Period A Placebo and ADT (8 Weeks) | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment) | Period A+ Placebo and ADT (Non-randomised Patients)
Started | 0 | 442 | 444 | 770
Completed | 0 | 380 | 349 | 653
Not Completed | 0 | 62 | 95 | 117
Not completed — Adverse Event | 0 | 13 | 27 | 16
Not completed — Lack of Efficacy | 0 | 9 | 11 | 6
Not completed — Withdrawal by Subject | 0 | 28 | 35 | 47
Not completed — Protocol Violation | 0 | 1 | 4 | 6
Not completed — Non-compliance with IMP | 0 | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 2 | 5 | 11
Not completed — Withdrawal before treatment | 0 | 1 | 0 | 0
Not completed — Administrative or other reasons | 0 | 6 | 10 | 28

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Patients: Period A
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 1986
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1402
  Male | 584
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 1918
  More than one race | 0
  Unknown or Not Reported | 46
Region of Enrollment [Number; unit: participants]
  Russian Federation | 121
  Romania | 15
  United States | 78
  Ukraine | 189
  United Kingdom | 168
  Canada | 30
  Latvia | 84
  Sweden | 85
  Finland | 136
  Poland | 325
  Mexico | 72
  Bulgaria | 119
  Lithuania | 76
  Germany | 325
  Estonia | 161
  Korea, Republic of | 2

OUTCOME MEASURES:

1. Primary Outcome: Full Remission During the Randomised Treatment Period
Description: Full remission is defined as a Montomery and Åsberg Depression Rating Scale (MADRS) total score ≤10 and a ≥50% decrease from randomisation in MADRS total score for at least 8 consecutive weeks during randomized treatment. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). The MADRS total score is the sum of the 10 items.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Number; unit: participants
Groups:
- Period B Placebo and ADT (24 Weeks Randomised Treatment): Placebo adjunct to open-label treatment with a commercially available ADT
  Placebo: Once daily, tablets, orally
- Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment): Brexpiprazole adjunct to open-label treatment with a commercially available ADT
  Brexpiprazole: 1, 2, or 3 mg/day, once daily dose, tablets, orally
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 441 | 444
participants | 110 | 95
Statistical Analysis 1: Comparison: Period B Placebo and ADT (24 Weeks Randomised Treatment) vs Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment); Test type: Superiority; p = 0.2641, Regression, Logistic; Model included MADRS total score at the randomisation visit, treatment group, country, and the randomisation criteria used; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.60 to 1.15]

2. Secondary Outcome: Full Functional Remission During the Randomised Treatment Period
Description: Full functional remission is defined as a Sheehan Disability Scale (SDS) total score <=6 and all SDS domain scores <=2 observed for at least 8 consecutive weeks during the randomised treatment period. The SDS assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 441 | 444
participants | 73 | 68

3. Secondary Outcome: Full Global Score Remission During the Randomised Treatment Period
Description: Full global score remission is defined as a Clinical Global Impression - Severity of Illness (CGI-S) score <=2 observed for at least 8 consecutive weeks during the randomised treatment period. The CGI-S is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis, on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 441 | 444
participants | 143 | 121

4. Secondary Outcome: Total Time in Remission During the Randomised Treatment Period
Description: The total time the patient spends in remission during randomised treatment. Remission is defined as a MADRS total score <=10 and a >=50% decrease from randomisation in MADRS total score. Time in remission is defined as the sum of days over all periods between Period B visits where remission was obtained. The period between two visits is counted as in remission if the patient was in remission when the period started.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 441 | 444
Number of days | 33.5 (46.1) | 30.0 (44.3)

5. Secondary Outcome: Time to Full Remission During the Randomised Treatment Period
Description: The time from randomisation until full remission has been obtained. Full remission is defined as a MADRS total score ≤10 and a ≥50% decrease from randomisation in MADRS total score for at least 8 consecutive weeks during randomised treatment. The time to full remission was calculated using Kaplan-Meier Methods.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 441 | 444
Days | NA [NA to NA] — The median number of days to full remission was not estimable (less than 50% of the patients were in full remission). | NA [NA to NA] — The median number of days to full remission was not estimable (less than 50% of the patients were in full remission).

6. Secondary Outcome: Full Remission Sustained During the Randomised Treatment Period
Description: Full remission sustained is defined as having obtained full remission and remain in remission until completion of the study. Full remission is defined as a MADRS total score ≤10 and a ≥50% decrease from randomisation in MADRS total score for at least 8 consecutive weeks during randomised treatment.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 441 | 444
participants | 105 | 84

7. Secondary Outcome: Change From Randomisation to Week 6 in MADRS Total Score During the Randomised Treatment Period
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). The MADRS total score is the sum of the 10 items.
Time Frame: From randomisation to week 6
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 422 | 422
units on a scale | -5.9 (0.4) | -6.3 (0.4)

8. Secondary Outcome: Change From Randomisation to Week 24 in MADRS Total Score During the Randomised Treatment Period
Description: as for outcome 7
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 361 | 333
Units on a scale | -12.6 (0.6) | -11.5 (0.6)

9. Secondary Outcome: Response at Week 6 During the Randomised Treatment Period
Description: Response is defined as a >=50% decrease from randomisation in MADRS total score.
Time Frame: From randomisation to week 6
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B. Last Observation Carried Forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 440 | 442
participants | 76 | 82

10. Secondary Outcome: Response at Week 24 During the Randomised Treatment Period
Description: Response is defined as a >=50% decrease from randomisation in MADRS total score.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 440 | 442
participants | 236 | 223

11. Secondary Outcome: Remission at Week 6 During the Randomised Treatment Period
Description: Remission is defined as a MADRS total score <=10 and a >=50% decrease from randomisation in MADRS total score.
Time Frame: From randomisation to week 6
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 440 | 442
participants | 46 | 53

12. Secondary Outcome: Remission at Week 24 in the Randomised Treatment Period
Description: Remission is defined as a MADRS total score <=10 and a >=50% decrease from randomisation in MADRS total score.
Time Frame: From randomisation to end of Period B (24 weeks)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 440 | 442
participants | 198 | 176

13. Secondary Outcome: Change From Randomisation to Week 6 in SDS Total Score During the Randomised Treatment Period
Description: The SDS assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment.
Time Frame: From randomisation to week 6
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 422 | 421
units on a scale | -3.0 (0.3) | -2.9 (0.3)

14. Secondary Outcome: Change From Randomisation to Week 24 in SDS Total Score During the Randomised Treatment Period
Description: as for outcome 13
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 361 | 333
units on a scale | -6.7 (0.5) | -5.5 (0.5)

15. Secondary Outcome: Change From Randomisation to Week 6 in CGI-S Score During the Randomised Treatment Period
Description: The CGI-S is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: From randomisation to week 6
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 422 | 422
units on a scale | -0.8 (0.1) | -0.8 (0.1)

16. Secondary Outcome: Change From Randomisation to Week 24 in CGI-S Score During the Randomised Treatment Period
Description: as for outcome 15
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 361 | 333
units on a scale | -1.7 (0.1) | -1.5 (0.1)

17. Secondary Outcome: Change From Randomisation to Week 6 in Q-LES-Q (SF) Total Score During the Randomised Treatment Period
Description: The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. The Q-LES-Q short form (SF) contains 16 items from the general activities section. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good). The total score is the sum of the first 14 items. The last two scores are stand-alone items. The total score ranges from 14 to 70.
Time Frame: From randomisation to week 6
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 422 | 421
units on a scale | 3.5 (0.4) | 3.2 (0.4)

18. Secondary Outcome: Change From Randomisation to Week 24 in Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q (SF)) Total Score During the Randomised Treatment Period
Description: as for outcome 17
Time Frame: From randomisation to end of Period B (24 weeks)
Population: All randomised patients who took at least one dose of randomised treatment (brexpiprazole or placebo) in Period B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Period B Placebo and ADT (24 Weeks Randomised Treatment) | Period B Brexpiprazole and ADT (24 Weeks Randomised Treatment)
Number analyzed (Participants) | 361 | 333
units on a scale | 7.7 (0.7) | 6.2 (0.7)

ADVERSE EVENTS:
Time Frame: Randomisation to end of study (28 weeks)
Description: Treatment-Emergent Adverse Events are reported in this section
Groups:
- Placebo and ADT: Placebo adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Placebo: Once daily, tablets, orally
- Brexpiprazole and ADT: Brexpiprazole adjunct to open-label treatment with a commercially available ADT
  Brexpiprazole: 1, 2, 3, mg/day, once daily, tablets, orally
Arm/Group | Placebo and ADT | Brexpiprazole and ADT
Serious Adverse Events (participants affected / at risk) | 13/441 | 9/444
Other Adverse Events (participants affected / at risk) | 97/441 | 108/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo and ADT (N=441) | Brexpiprazole and ADT (N=444)
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
False positive investigation result (Investigations) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 1
Self injurious behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1/302 | 0/307
Family stress (Social circumstances) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo and ADT (N=441) | Brexpiprazole and ADT (N=444)
Nasopharyngitis (Infections and infestations) | 34 | 28
Accidental overdose (Injury, poisoning and procedural complications) | 25 | 27
Weight increased (Investigations) | 22 | 42
Headache (Nervous system disorders) | 31 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No